CLINICAL TRIAL: NCT00660530
Title: An Evaluation of Chewed vs. Crushed Lanthanum Carbonate in the Efficacy of Phosphate Binding in Hemodialysis Patients
Brief Title: Chewed vs. Crushed Lanthanum Carbonate in Hemodialysis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Shire (Industry)
Responsible Party: Principal Investigator, Alan Lau, Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0588
Record Dates: First submitted 2008-04-09; First posted 2008-04-17 (Estimated); Results first posted 2020-10-01 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Hyperphosphatemia; Kidney Disease
Keywords: stage 5; chronic; hemodialysis
MeSH Terms: conditions — Hyperphosphatemia; Kidney Diseases; Bronchiolitis Obliterans Syndrome | interventions — lanthanum carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): One week before the administration of crushed or chewed lanthanum, the subjects were instructed to discontinue their P-binding agents, if prescribed previously. At the end of the 1-week washout period, subjects whose serum P exceeded 5.5 mg/dL were randomized to receive, in a crossover fashion, lanthanum 1000 mg (Fosrenol, Shire US Inc., Wayne, PA, USA) 3 times daily to be chewed with meals (chewed LAN) or lanthanum 1000 mg crushed into a ﬁne powder and taken with meals 3 times daily (crushed LAN), for 4 weeks each. The lanthanum tablets were crushed into a ﬁne powder using a mortar and pestle by the investigators, individually wrapped in powder packets and dispensed to the subjects on a weekly basis. The subjects were instructed to empty the powder into a small plastic cup provided, mix with 2 tablespoonfuls of applesauce and take it with meals. After each treatment (chewed or crushed LAN), there was a 1-week washout period.
  Interventions: Drug: Lanthanum Carbonate Chewable Product
- 2 (Experimental): After the one-week washout period, the subject received the other lanthanum treatment (chewed or crushed) that they did not receive in the initial treatment period.
  Interventions: Drug: Lanthanum carbonate crushed powder

INTERVENTIONS:
Drug: Lanthanum Carbonate Chewable Product — Lanthanum carbonate 1 g to be chewed, three times daily with meals
  Other Names: Fosrenol
  Arms: 1
Drug: Lanthanum carbonate crushed powder — Lanthanum carbonate (Fosrenol) 1 g crushed into a fine powder, three times daily with meal
  Other Names: Fosrenol
  Arms: 2

SUMMARY:
Patients with end-stage renal disease (ESRD) commonly develop hyperphosphatemia due to the loss of excretory function of the kidney. This in turn may lead to the development of secondary hyperparathyroidism (SHPT) and renal osteodystrophy. Lanthanum carbonate, a phosphate binding agent, works by releasing lanthanum ions in the gastrointestinal tract to bind dietary phosphate and is effective in the management of hyperphosphatemia and in preventing secondary hyperparathyroidism.

Patients taking lanthanum carbonate as part of their phosphate binder therapy are counseled to chew the tablets completely before swallowing, with or immediately after meals. However, ESRD patients who are intubated or are receiving enteral tube feedings are unable to chew the lanthanum carbonate tablets. For such patients, medications are commonly crushed and administered through a gastrostomy tube (G-tube). Some patients may also prefer to crush the lanthanum carbonate tablets and mix it with food instead of chewing. To date, it is not known if crushing the lanthanum carbonate tablets prior to administration and taking it with food will be as efficacious as chewing it.

The objective of this study is to compare the efficacy of phosphate binding between chewed and crushed lanthanum carbonate in patients undergoing hemodialysis.

DETAILED DESCRIPTION:
Study subjects Men and women at least 18 years of age, receiving HD for at least 3 months, with serum P concentrations 45.5 mg/dL at the end of the washout period, and on a stable dose of P binder and/or active vitamin D (if prescribed previously) for at least 1 month before the study were eligible for study participation. Patients were excluded if they did not respond to P binder therapy previously, had a known noncompliance with oral medications (e.g., failure to ﬁll a prescription or to take medications as prescribed), severe hyperparathyroidism deﬁned as intact-PTH (i-PTH) 4500 pg/mL, were taking any calcium (Ca)-, magnesium-, or aluminum-containing antacids or used an investigational agent within 30 days of study entry.

Study design This study was approved by the University of Illinois at Chicago Institutional Review Board. Informed consent was obtained from the subjects before any study procedures were initiated. One week before the administration of crushed or chewed lanthanum, the subjects were in-structed to discontinue their P-binding agents (calcium carbonate, calcium acetate, sevelamer hydrochloride, and/or lanthanum carbonate), if prescribed previously. At the end of the 1-week washout period, subjects whose serum P exceeded 5.5 mg/dL were randomized to receive, in a crossover fashion, lanthanum 1000 mg (Fosrenol, Shire US Inc., Wayne, PA, USA) 3 times daily to be chewed with meals (chewed LAN) or lanthanum 1000 mg crushed into a ﬁne powder and taken with meals 3 times daily (crushed LAN), for 4 weeks each. The lanthanum tablets were crushed into a ﬁne powder using a mortar and pestle by the investigators, individually wrapped in powder packets and dispensed to the subjects on a weekly basis. The subjects were instructed to empty the powder into a small plastic cup provided, mix with 2 tablespoonfuls of applesauce and take it with meals. After each treatment (chewed or crushed LAN), there was a 1-week washout period.

Throughout the course of the study, the subjects were asked to keep a constant dietary P intake. In addition, each subject was provided with a dietary log for recording their daily dietary intake.

Sample collection and study endpoints Blood samples were collected at the end of each washout period (baseline) and weekly (weeks 1-4) during lanthanum treatment for the determination of serum P, Ca, i-PTH, and albumin (alb) concentrations. Changes in serum P from baseline for crushed and chewed lanthanum were compared. In addition, the study subjects were asked to complete a questionnaire to assess the presence of any study-related adverse events at the end of each treatment arm.

Statistical considerations Assuming a coefﬁcient variation of 15% to 25% for serum P concentrations, a sample size of 11 to 15 was estimated to provide at least 80% power to detect a 25% difference in serum P between study treatments, using a 2-sided test and a of 0.05. Statistical analyses were performed using PASW (SPSS), version 17.0 (Chicago, IL, USA). Descriptive statistics were used to report all results. The changes in serum P, Ca, i-PTH, and alb were compared between the 2 treatment arms using paired sample t test. A P value <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years of age or older
* Have been on hemodialysis for at least 3 months
* Women of child-bearing potential (premenopausal and not surgically sterilized) who have a negative serum pregnancy test
* On a stable dose of phosphate binder for at least 1 month prior to the study
* On a stable dose of active vitamin D (if previously prescribed) for at least 1 month prior to the study
* Serum phosphorus concentrations > 5.5 mg/dL (1.78 mmol/L) at the end of the washout period

Exclusion Criteria:

* Did not previously respond to phosphate binder therapy
* Known non-compliance with oral medications
* Severe hyperparathyroidism defined as intact-PTH (i-PTH) > 500 pg/ml
* Taking any calcium-, magnesium- or aluminum-containing antacids
* Use of an investigational agent within 30 days of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-01; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan H Lau, Pharm.D., Principal Investigator — Univsersity of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Men and women at least 18 years of age, receiving hemodialysis (HD) for at least 3 months, with serum P concentrations > 5.5 mg/dL at the end of the washout period, and on a stable dose of P binder and/or active vitamin D (if previously prescribed) for at least 1 month prior to the study were eligible for study participation.
Pre-assignment Details: Patients were excluded if they did not previously respond to P binder therapy, had a known non-compliance with oral medications, severe hyperparathyroidism defined as intact-PTH (i-PTH) > 500 pg/ml, were taking any calcium-, magnesium- or aluminum-containing antacids or used an investigational agent within 30 days of study entry.
Groups:
- Chewed or Crushed Lanthanum Carbonate: Lanthanum carbonate 1 g to be chewed or crushed, three times daily with meals, after 1-week washout period, then Lanthanum carbonate 1 g to be chewed crushed, three times daily with meals (the treatment that the subject did not receive in the initial treatment).
Period: Overall Study
Arm/Group | Chewed or Crushed Lanthanum Carbonate
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Chewed or Crushed Lanthanum Carbonate: Lanthanum carbonate 1 g to be chewed or crushed, three times daily with meals
Arm/Group | Chewed or Crushed Lanthanum Carbonate
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Serum Phosphorous Concentration
Description: measure of serum P concentration
Time Frame: Week 1-4 mean
Measure: Mean (Standard Error); unit: mg/dL
Groups:
- Chewed Lanthanum Carbonate: Lanthanum carbonate 1 g to be chewed, three times daily with meals
- Crushed Lanthanum Carbonate: Lanthanum carbonate 1 g crushed into a fine powder, three times daily with meal
  Lanthanum carbonate: Lanthanum carbonate 1 g crushed into a fine powder, three times daily with meal
Arm/Group | Chewed Lanthanum Carbonate | Crushed Lanthanum Carbonate
Number analyzed (Participants) | 11 | 11
mg/dL | 2.0 (0.5) | 1.7 (0.4)

ADVERSE EVENTS:
Time Frame: 4 weeks for each cross-over period
Description: non-systematic assessment
Groups:
- Crushed Lanthanum Carbonate: Lanthanum carbonate 1 g crushed into a fine powder, three times daily with meal
Arm/Group | Chewed Lanthanum Carbonate | Crushed Lanthanum Carbonate
Serious Adverse Events (participants affected / at risk) | 1/11 | 2/11
Other Adverse Events (participants affected / at risk) | 7/11 | 6/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chewed Lanthanum Carbonate (N=11) | Crushed Lanthanum Carbonate (N=11)
Severe Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Severe Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chewed Lanthanum Carbonate (N=11) | Crushed Lanthanum Carbonate (N=11)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dizziness (Vascular disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No